CLINICAL TRIAL: NCT05248529
Title: Effect of Preoperative Education Based on Roy Adaptation Model in Patients With Hip or Knee Arthroplasty on Physical Adaptation and Mobility
Brief Title: Effect of Preoperative Education Based on Roy Adaptation Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Merve Ozsoy Durmaz, MSc, Research Assistant, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: mozsoy
Record Dates: First submitted 2022-01-24; First posted 2022-02-21 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Orthopedic Disorder
Keywords: Roy Adaptation Model; hip arthroplasty; knee arthroplasty; physical adaptation; preoperative education
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: The sample was composed of 78 individuals 41 experimental and 37 control. The intervention group was given practical training in accordance with the adaptation booklet prepared by the researcher. Patients' physical adaptation and mobility were evaluated using the Patient Mobility Scale and Observer Mobility Scale and Physical Adaptation Assesment Form. Data of the control and intervention groups were collected two times: preoperative and within 12 hours before the discharge.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Within 12-24 hours before the surgery, the demonstrative education was given based on 'Hip Replacement Adaptation Booklet' and 'Knee Replacement Adaptation Booklet' to the patients in the intervention group.
  Interventions: Other: Education booklet
- Control gorup (No Intervention): Routine preoperative preparation training was performed to the patients in the control group.

INTERVENTIONS:
Other: Education booklet — Hip/Knee Replacement Adaptation Booklet explains preoperative preparation, post-operative care practices, how to walk with walker, what needs to be done at home after discharge
  Arms: Intervention group

SUMMARY:
This research was conducted as a randomized controlled experiment to determine the effect of the education given by the Physiological Mode of Roy Adaptation Model in patients with hip or knee arthroplasty on physical adaptation and mobility.

DETAILED DESCRIPTION:
The research was conducted between 01.11.2017 - 01.04.2018 at the Orthopedics and Traumatology Surgery Service of a private University Hospital in Istanbul.

In the study, the number of samples to be taken; the training, the training group control group mobility scale scores between The Observer at least 5% of the study considering that would make a difference, and power 80%, α=0.05 and power analysis adopted by participants for each group were calculated and it was determined that there should be at least 27.

The sample was composed of 78 individuals 41 experimental and 37 control. Patients' physical adaptation and mobility were evaluated using the Patient Mobility Scale and Observer Mobility Scale and Physical Adaptation Assessment Form.

Randomization of the study was achieved by planning patients who met the inclusion and non-inclusion criteria for training and control groups sequentially, without dividing them into hip or knee arthroplasty. In the randomization table, those with the number 1 are assigned to the training group.

ELIGIBILITY:
Inclusion Criteria:

can read and write in Turkish A sufficient level of education to understand study procedures and training

Exclusion Criteria:

hospitalized due to fracture mental disability neurological disease undergone the same operation before received similar training before

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Weight | 5 days
  weight in kilograms. It was used to determine the body mass index.
height | 5 days
  height in meters. it was used to determine the body mass index.
Body Mass Index | 5 days
  Body Mass Index is a simple calculation using a person's height and weight. The formula is BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared.
Systolic and diastolic blood pressure | 5 days
  Both systolic and diastolic blood pressure is measured in units of millimeters of mercury (mmHg). It was used to determine the blood pressure of patients before mobilization.

SECONDARY OUTCOMES:
The Observer Mobility Scale | 5 days
  1 point indicates that the activity can be performed independently without verbal warning and physical assistance, 5 points indicate that the patient cannot perform the activity independently despite the verbal warning and physical assistance. The lowest score that can be obtained from the scale is 4 and the highest score is 20.
The Patient Mobility Scale | 5 days
  As a scale score, 1 indicates that the patient has no pain during the activity and the level of difficulty when moving is minimal, while 5 indicates that the patient's pain during the activity is unbearable and the level of difficulty is greatest. The lowest score that can be obtained from the scale is 8 and the highest score is 40.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Ozsoy Durmaz, Study Director — Medipol University
Locations (1):
- Yeditepe University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
An application for publication will be submitted in 2022.
Supporting Information: CSR
Time Frame: 6 months
Access Criteria: studies on hip and knee arthroplasty